CLINICAL TRIAL: NCT07154251
Title: Utilizing a Community Health Worker in the Role of a Diabetes Technology Coach for Black Children Using Automated Insulin Delivery and Not Meeting Glycemic Targets (CHWs AID Youth)
Brief Title: Utilizing Community Health Workers as Diabetes Technology Coaches for Children With Type 1 Diabetes Using Automated Insulin Delivery
Acronym: CHWs AID Youth
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Sarah A. MacLeish, Associate Professor of Pediatrics, University Hospitals Cleveland Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY20250042
Record Dates: First submitted 2025-08-26; First posted 2025-09-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Type 1 Diabetes (T1D)
Keywords: Automated insulin delivery; Community Health Worker; Disparities; Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Community Health Workers

STUDY DESIGN:
Intervention Model Description: Single arm pilot intervention study with use of historic controls
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Community Health Worker (Experimental): Community Health Workers will meet with families monthly in the role of a diabetes technology coach, with additional visits as needed.
  Interventions: Other: Community Health Worker

INTERVENTIONS:
Other: Community Health Worker — Community Health Worker will meet with families monthly (and more often as needed) in the role of a diabetes technology coach

SUMMARY:
This study uses community health workers (CHW) as diabetes technology coaches for African American children using automated insulin delivery systems but have an HbA1c of 8% or higher. Families will meet with the CHW monthly x 6 months with additional visits as needed. All participants and parents/guardians will fill out questionnaires at the beginning and end of the 6 month intervention in addition to an interview at 6 months. This will be followed by 6 months with no extra help from the CHW, but we will continue to follow CGM and pump download data.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported as non-Hispanic Black
* Clinical diagnosis of type 1 diabetes, requiring treatment with insulin at the time of consent
* Currently using, or have used within the past 3 months, an automated insulin delivery system (consisting of a continuous glucose monitor and an insulin pump as well as an automated insulin delivery algorithm)
* Clinical care provided at UH Cleveland Medical Center
* Has not previously worked with a community health worker for help with diabetes technology

Exclusion Criteria:

* Clinical diagnosis of Type 2 or monogenic diabetes
* Completed high school
* At least 1 parent/guardian or family support person not willing to participate
* Non-English speaking guardians
* Has not used automated insulin delivery within the past 3 months
* Has previously worked with a CHW for help with diabetes technology
* Custody of children and family services

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Estimated)
Dates: Start 2025-11-06 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in capillary HbA1c | Baseline, 3 months, 6 months, 9 months, 12 months
Change in number of participants who use an automated insulin delivery system with at least 80% time in automated mode over the past 30 days, as measured by download of data from the automated insulin delivery system | Baseline, 3 months, 6 months, 9 months, 12 months

SECONDARY OUTCOMES:
Change in time in range (70-180 mg/dL) as measured by continuous glucose monitoring | Baseline, 3 months, 6 months, 9 months, 12 months
  Time in range (70-180 mg/dL) will be assessed over the 30 day increment prior to each study visit
Change in time under 70 mg/dL as measured by continuous glucose monitoring | Baseline, 3 months, 6 months, 9 months, 12 months
  Time under 70 mg/dL will be assessed over the 30 day time increment prior to each study visit
Change in time over 250 mg/dL as measured by continuous glucose monitoring | Baseline, 3 months, 6 months, 9 months, 12 months
  Time above 250 mg/dL will be assessed over the 30 day increment prior to each study visit
Change in continuous glucose monitor wear time as measured by continuous glucose monitoring | Baseline, 3 months, 6 months, 9 months, 12 months
  Wear time will be assessed over the 30 day increment prior to each study visit
Change in time in automated mode as measured by automated insulin delivery system | Baseline, 3 months, 6 months, 9 months, 12 months
  Time in automated mode will be assessed over the 30 day increment prior to each study visit.
Change in psychosocial functioning of children/adolescents, as measured by the strengths and difficulties questionnaire given to parents/guardians | Baseline, 6 months
  Description: 25-item questionnaire using a 3-point Likert scale, with one being not true and 3 being certainly
Change in diabetes family conflict, as measured by the Diabetes Family Conflict Scale | Baseline, 6 months
  19-item questionnaire using 3-point Likert scale, where 1 is almost never and 3 is almost always
Change in child/adolescent quality of life, as measured by PedsQL Type 1 diabetes module by parent-proxy | Baseline, 6 months
  28-item questionnaire using 5-point Likert scale, where 0 is almost never a problem and 4 is almost always a problem
Change in parental burden related to diabetes, as measured by Problem Areas in Pediatric Diabetes - Parent Revised Version | Baseline, 6 months
  18-item questionnaire using 5-point Likert scale, where 0 is agree and 4 is disagree
Change in medical distrust, as measured by the Group Based Medical Distrust Scale | Baseline, 6 months
  12-item questionnaire using 5 point Likert scale, where 1 is strongly disagree and 5 is strongly agree
Change personal frequency of discrimination in healthcare, as measured by the Racism in Healthcare Index | Baseline, 6 months
  7-item questionnaire regarding frequency of discrimination in healthcare ranging from never to 4 times or more in a lifetime
Change in perceptions of racism in healthcare, as measured by the Racism in Healthcare Index | Baseline, 6 months
  4-item questionnaire using 5 point Likert scale where 1 is strongly disagree and 5 is strongly agree
Change in diabetes specific attitudes towards technology as measured by the Diabetes Specific Technology Attitudes Scale | Baseline, 6 months
  5-item questionnaire using 5 point Likert scale, where 1 is strongly disagree and 5 is strongly agree
Change in barriers to technology as measured by Barriers to Technology Checklist | Baseline, 6 months
  19-item yes/no questionnaire
Change in diabetes management self-efficacy as measured by the Self-Efficacy for Diabetes Self-Management scale short version | Baseline, 6 months
  10-item questionnaire using 6-point Likert scale, where 1 is "very sure I can't" and 6 is "very sure I can"
Change in Benefits and Burdens of CGM as measured by Benefits and Burdens of CGM scale | Baseline, 6 months
  16-item questionnaire using 5-point Likert scale, where 1 is strongly disagree and 5 is strongly agree
Episodes of Diabetic Ketoacidosis as measured by chart review | up to 12 months
  DKA defined as presence of all of the following: 1) blood glucose greater than 250 mg/dL, 2) pH less than 7.3 OR bicarbonate less 15 mEq/L, 3)Moderate or large ketones in urine OR blood ketone >3 mmol/L, 4) Requiring treatment within a health care facility.
Episodes of severe hypoglycemia as measured by chart review | Up to 12 months
  Unconscious or having a seizure due to hypoglycemia

OTHER OUTCOMES:
Number of meetings with community health worker | Up to 6 months
Duration in hours/minutes of meetings with community health worker | Up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sarah A MacLeish, DO, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
This is a pilot study